CLINICAL TRIAL: NCT04932122
Title: Outcomes of Surgical Excision of Dorsal Wrist Ganglia With or Without Partial Wrist Denervation
Brief Title: Outcomes After Dorsal Wrist Ganglia Excision With or Without PIN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study recruitment stopped due to recruitment problems
Sponsor: Kenneth Taylor, M.D. (Other)
Responsible Party: Sponsor-Investigator, Kenneth Taylor, M.D., Professor of Orthopaedics and Rehabilitation, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00016888
Record Dates: First submitted 2021-05-24; First posted 2021-06-18 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Wrist Ganglion; Ganglion Cysts; Hand Ganglion; Denervation Atrophy
Keywords: ganglion cysts; dorsal wrist ganglia; neurectomy; denervation; posterior interosseous nerve
MeSH Terms: conditions — Ganglion Cysts

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the study team member who is performing the physical exam (including range of motion and grip/pinch strength testing) will be blinded to the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dorsal wrist ganglion alone (DWG) (Active Comparator): Dorsal wrist ganglion excision alone
  Interventions: Procedure: Dorsal wrist ganglion alone (DWG)
- DWG with PIN (Active Comparator): Dorsal wrist ganglion excision with posterior interosseus neurectomy (PIN)
  Interventions: Procedure: DWG/PIN

INTERVENTIONS:
Procedure: Dorsal wrist ganglion alone (DWG) — Patients assigned to this arm will undergo dorsal wrist ganglion cyst excision alone.
  Arms: Dorsal wrist ganglion alone (DWG)
Procedure: DWG/PIN — Patients assigned to this arm will undergo dorsal wrist ganglion excision and the addition of a partial wrist denervation by resecting the common terminal sensory branch of the posterior interosseus nerve (PIN)..
  Arms: DWG with PIN

SUMMARY:
The purpose of this study is to determine if a statistical significance exists between outcomes of patients treated for dorsal wrist ganglion cyst with excision alone versus excision and the addition of a partial wrist denervation by resecting the common terminal sensory branch of the PIN (posterior interosseus nerve). Our hypothesis is that addition of PIN improves outcome after dorsal wrist ganglion excision as indicated by post-operative pain, function, ability to perform activities of daily living, and physical exam findings.

DETAILED DESCRIPTION:
The primary endpoint will be outcomes on subject surveys and questionnaires. Data will be collected pre- and post-operatively at 2 weeks, 12 weeks, 6 months, and one year. Four questionnaires will be used, including the Visual Analog Pain Score (VAS), Disabilities of the Arm, Shoulder, and Hand (QuickDASH) questionnaire, as well as the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference (PI), and the PROMIS Pain Behavior (PB) questionnaires.

Secondary outcomes include physical examination consisting of pre- and post-operative pinch and grip strength testing, and active range of motion including wrist flexion and extension ulnar and radial deviation, and weight bearing extension. These will be performed at 2 weeks, 12 weeks, and 6 months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age
* Gender: male/female (non-pregnant)
* Diagnosis of symptomatic (pain and limited ability to perform activities of daily living) dorsal wrist ganglion cyst
* Subjects who have chosen surgical management for their ganglion cyst diagnosis
* Fluent in written and spoken English
* Subject is able to provide voluntary, written informed consent
* Subject, in the opinion of the clinical investigator, is able to understand the clinical investigation and is willing to perform all study procedures and follow-up visits
* Non-Prisoners

Exclusion Criteria:

* Less than 18 years of age
* Non-elective surgery for this diagnosis
* Chronic wrist instability of the operative extremity
* Comorbid neurologic maladies of the operative extremity
* Prior wrist surgery on either extremity
* Non-English speaking
* Prisoners
* Pregnancy
* Cognitive Impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2026-02-03 (Actual); Study Completion 2026-02-03 (Actual)

PRIMARY OUTCOMES:
Pain measured with the Visual Analog Pain Scale (VAS) | Preop to One Year Post-Op
  Self-report measurement that assesses a person's perceived level of pain
Physical Function measured with the Disabilities of the Arm, Shoulder and Hand questionnaire (QuickDASH) | Preop to One Year Post-Op
  11-Item questionnaire that measures physical function and symptoms in people with musculoskeletal disorders of the upper limb
Pain interference measured with the Patient-Reported Outcomes Measurement Information (PROMIS) Pain Interference instrument | Preop to One Year Post-Op
  This instrument measures the self-reported consequences of pain on relevant aspects of one's life and may include the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities.
Pain behavior measured with the Patient-Reported Outcomes Measurement Information (PROMIS) Pain Behavior instrument | Preop to One Year Post-Op
  This instrument measures self-reported external manifestations of pain: behaviors that typically indicate to others that an individual is experiencing pain.

SECONDARY OUTCOMES:
Change in strength utilizing hand grip measurements | Preop to 6 Months Post-Op
  This measurement provides information about muscle strength health in the hand and forearms. The average of three measurements is taken using a hand-held dynamometer
Change in strength utilizing finger lateral pinch measurements | Preop to 6 Months Post-Op
  This measurement provides information about the functional strength of one's pinching action of the hand using a mechanical pinch gauge. The average of three measurements will be taken at each time frame.
Change in strength utilizing finger tip pinch measurements | Preop to 6 Months Post-Op
  This measurement provides information about the functional strength of one's pinching action of the hand using a mechanical pinch gauge. The average of three measurements will be taken at each time frame.
Change in strength utilizing finger three-point pinch measurements | Preop to 6 Months Post-Op
  This measurement provides information about the functional strength of one's pinching action of the hand using a mechanical pinch gauge. The average of three measurements will be taken at each time frame.
Change in wrist flexion | Preop to 6 Months Post-Op
  This measurement indicates the range of motion of the wrist utilizing a goniometer
Change in wrist extension | Preop to 6 Months Post-Op
  This measurement indicates the range of motion of the wrist utilizing a goniometer
Change in wrist weight bearing extension | Preop to 6 Months Post-Op
  This measurement indicates the range of motion of the wrist utilizing a goniometer
Change in wrist ulnar deviation | Preop to 6 Months Post-Op
  This measurement indicates the range of motion of the wrist from side to side. This movement flexes the hand toward the ulnar bone in the arm. This is measured with a goniometer.
Change in wrist radial deviation | Preop to 6 Months Post-Op
  This measurement indicates the range of motion of the wrist from side to side. This movement flexes the hand toward the radial bone in the arm. This is measured with a goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Taylor, MD, Principal Investigator — Penn State Health Milton S Hershey Medical Center
Locations (2):
- United States (2):
  - Penn State Health Medical Group - Camp Hill Specialties, Camp Hill, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania

REFERENCES:
- [Background] Ho PC, Griffiths J, Lo WN, Yen CH, Hung LK. Current treatment of ganglion of the wrist. Hand Surg. 2001 Jul;6(1):49-58. doi: 10.1142/s0218810401000540. PMID 11677666
- [Background] Thornburg LE. Ganglions of the hand and wrist. J Am Acad Orthop Surg. 1999 Jul-Aug;7(4):231-8. doi: 10.5435/00124635-199907000-00003. PMID 10434077
- [Background] Angelides AC, Wallace PF. The dorsal ganglion of the wrist: its pathogenesis, gross and microscopic anatomy, and surgical treatment. J Hand Surg Am. 1976 Nov;1(3):228-35. doi: 10.1016/s0363-5023(76)80042-1. PMID 1018091
- [Background] Clay NR, Clement DA. The treatment of dorsal wrist ganglia by radical excision. J Hand Surg Br. 1988 May;13(2):187-91. doi: 10.1016/0266-7681_88_90135-0. PMID 3385297
- [Background] Dellon AL, Seif SS. Anatomic dissections relating the posterior interosseous nerve to the carpus, and the etiology of dorsal wrist ganglion pain. J Hand Surg Am. 1978 Jul;3(4):326-32. doi: 10.1016/s0363-5023(78)80032-x. PMID 681715
- [Background] Carr D, Davis P. Distal posterior interosseous nerve syndrome. J Hand Surg Am. 1985 Nov;10(6 Pt 1):873-8. doi: 10.1016/s0363-5023(85)80165-9. PMID 4078272
- [Background] Dellon AL. Partial dorsal wrist denervation: resection of the distal posterior interosseous nerve. J Hand Surg Am. 1985 Jul;10(4):527-33. doi: 10.1016/s0363-5023(85)80077-0. PMID 4020064
- [Background] Faithfull DK, Seeto BG. The simple wrist ganglion--more than a minor surgical procedure? Hand Surg. 2000 Dec;5(2):139-43. doi: 10.1142/s0218810400000235. PMID 11301508
- [Background] Fukumoto K, Kojima T, Kinoshita Y, Koda M. An anatomic study of the innervation of the wrist joint and Wilhelm's technique for denervation. J Hand Surg Am. 1993 May;18(3):484-9. doi: 10.1016/0363-5023(93)90096-L. PMID 8515020
- [Background] Hudak PL, Amadio PC, Bombardier C. Development of an upper extremity outcome measure: the DASH (disabilities of the arm, shoulder and hand) [corrected]. The Upper Extremity Collaborative Group (UECG). Am J Ind Med. 1996 Jun;29(6):602-8. doi: 10.1002/(SICI)1097-0274(199606)29:63.0.CO;2-L. PMID 8773720
- [Background] Chung KC, Pillsbury MS, Walters MR, Hayward RA. Reliability and validity testing of the Michigan Hand Outcomes Questionnaire. J Hand Surg Am. 1998 Jul;23(4):575-87. doi: 10.1016/S0363-5023(98)80042-7. PMID 9708370
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Szabo RM. Outcomes assessment in hand surgery: when are they meaningful? J Hand Surg Am. 2001 Nov;26(6):993-1002. doi: 10.1053/jhsu.2001.29487. PMID 11721242
- [Background] Gundes H, Cirpici Y, Sarlak A, Muezzinoglu S. Prognosis of wrist ganglion operations. Acta Orthop Belg. 2000 Oct;66(4):363-7. PMID 11103488
- [Background] BUTLER ED, HAMILL JP, SEIPEL RS, DE LORIMIER AA. Tumors of the hand. A ten-year survey and report of 437 cases. Am J Surg. 1960 Aug;100:293-302. doi: 10.1016/0002-9610(60)90302-0. No abstract available. PMID 13806476
- [Background] Gummesson C, Atroshi I, Ekdahl C. The disabilities of the arm, shoulder and hand (DASH) outcome questionnaire: longitudinal construct validity and measuring self-rated health change after surgery. BMC Musculoskelet Disord. 2003 Jun 16;4:11. doi: 10.1186/1471-2474-4-11. Epub 2003 Jun 16. PMID 12809562
- [Background] Weinstein LP, Berger RA. Analgesic benefit, functional outcome, and patient satisfaction after partial wrist denervation. J Hand Surg Am. 2002 Sep;27(5):833-9. doi: 10.1053/jhsu.2002.35302. PMID 12239673
- [Background] Dell P. Benign, Aggressive, and Malignant Neoplasms. Hand Surgery Update, American Society for Surgery of the Hand, 1999, pg. 377.